CLINICAL TRIAL: NCT06032858
Title: Efficacy and Safety of Apremilast in Patients With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Efficacy and Safety of Apremilast in Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ghurki Trust and Teaching Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apremilast 30 mg twice daily (Experimental)
  Interventions: Drug: Apremilast 30mg

INTERVENTIONS:
Drug: Apremilast 30mg — Apremilast 30mg twice daily

SUMMARY:
Psoriasis is a long standing inflammatory, autoinflammatory disease linked with many comorbidities. Patients with moderate to severe plaque psoriasis can be managed with topical as well as systemic medications. FDA approved Apremilast as first drug to be taken orally in cases of psoriasis in mid 1990's. Currently, according to researchers best knowledge no study has been done on use of Apremilast in Pakistan. It has recently become available here. Keeping in view all the benefits of this drug, a study has been planned to check its effectiveness and safety 30mg twice a day, in patients with moderate to severe chronic plaque psoriasis based on Psoriasis area and severity index and Body surface area assessments in our population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed patients of chronic plaque psoriasis
* patients applicant for oral or parenteral treatments and for light therapy
* patients not responding to topical treatments

Exclusion Criteria:

* Patients who show hypersensitive reactions to apremilast to any of its inactive component
* Pregnancy
* Lactating mothers

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-06 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Psoriasis area and severity index | 16 weeks
body surface area | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Haroon Nabi, Study Director — Professor Department of Dermatology LMDC; Dr. Saira Muaaz, Principal Investigator — Department of Dermatology Ghurki Hospital; Dr. Hira Tariq, Study Chair — Senior Registrar Department of Dermatology Services Hospital; Dr. Sumera Hanif, Study Chair — Senior Registrar Department of Dermatology LMDC; Dr. Talat Akbar, Study Chair — Associate Professor, Dermatology, LMDC; Prof. Dr. Faria Asad, Study Chair — Head of Department Dermatology SIMS/ Services Hospital
Locations (1):
- Ghurki Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schafer P. Apremilast mechanism of action and application to psoriasis and psoriatic arthritis. Biochem Pharmacol. 2012 Jun 15;83(12):1583-90. doi: 10.1016/j.bcp.2012.01.001. Epub 2012 Jan 10. PMID 22257911
- [Background] Crowley J, Thaci D, Joly P, Peris K, Papp KA, Goncalves J, Day RM, Chen R, Shah K, Ferrandiz C, Cather JC. Long-term safety and tolerability of apremilast in patients with psoriasis: Pooled safety analysis for >/=156 weeks from 2 phase 3, randomized, controlled trials (ESTEEM 1 and 2). J Am Acad Dermatol. 2017 Aug;77(2):310-317.e1. doi: 10.1016/j.jaad.2017.01.052. Epub 2017 Apr 14. PMID 28416342